CLINICAL TRIAL: NCT00127036
Title: A Multicenter Trial for Microarray Analysis of Colon Cancer Outcome-A (MACCO-A)
Brief Title: Trial for Microarray Analysis of Colon Cancer Outcome-A (MACCO-A)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug now on market
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13449; R21 CA10135 (Other Grant/Funding Number: NCI); XEL390 (Other: Roche); 2005-0729 (Other: Pfizer)
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-12

CONDITIONS: Adenocarcinoma; Colon Cancer
Keywords: colon; adenocarcinoma; adenocarcinoma-colon; adenocarcinoma-rectum
MeSH Terms: conditions — Adenocarcinoma; Colonic Neoplasms; Rectal Neoplasms | interventions — XELOX; Oxaliplatin; Capecitabine; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XELOX + Bevacizumab (Experimental): Arm A: Anticipated 75 Patients - Drug: XELOX (which is Capecitabine + Oxaliplatin) by mouth + Bevacizumab intravenously as outlined in Intervention Description - To Disease Progression
  Interventions: Drug: XELOX; Drug: Bevacizumab
- XELIRI + Bevacizumab (Experimental): Arm B: Anticipated 75 Patients - Drug: XELIRI (which is Capecitabine + Irinotecan) by mouth + Bevacizumab intravenously as outlined in Intervention Description - To Disease Progression
  Interventions: Drug: XELIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: XELOX — XELOX: Oxaliplatin 130 mg/m^2 intravenously (IV); Capecitabine 825 mg/m^2 by mouth (po)
  Other Names: Oxaliplatin and Capecitabine
  Arms: XELOX + Bevacizumab
Drug: XELIRI — XELIRI: Irinotecan 240 mg/m^2 IV; Capecitabine 825 mg/m^2 by mouth (po)
  Other Names: Irinotecan and Capecitabine
  Arms: XELIRI + Bevacizumab
Drug: Bevacizumab — 7.5 mg/kg intravenously (IV)
  Other Names: Avastin®

SUMMARY:
The purpose of this study is to determine if the investigators can predict the sensitivity or resistance of colon cancer to the two available first line chemotherapy agents.

DETAILED DESCRIPTION:
Colorectal cancer is the third largest cause of cancer mortality in the United States. The treatment of metastatic colorectal cancer is undergoing rapid improvement. Currently, there are two major chemotherapy regimens, which can both be combined with anti-angiogenesis treatment. These regimens are 5-Fluorouracil (5-FU) + irinotecan and 5-FU + oxaliplatin. Each therapy has roughly similar rates of response, but it is unclear which specific therapy would benefit which patients. The advent of genome wide expression analysis provides a tool to analyze these differences. In the microarray analysis of colon cancer outcome trial, sponsored by the National Institutes of Health (NIH) and Moffitt Cancer Center, patients with newly diagnosed metastatic colon cancer are biopsied and samples are preserved in ribonucleic acid (RNA) later. Patients are then randomized to either one of two state of the art regimens: capecitabine + irinotecan + avastin (bevacizumab) or capecitabine + oxaliplatin + avastin. Response to chemotherapy, time to progression, and overall survival are end points of this trial. Once accrual of patients has been met, the investigators will compare genome wide expression patterns for each group.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients with metastatic, Response Evaluation Criteria In Solid Tumors (RECIST) measurable, adenocarcinoma of the colon and/or rectum are eligible provided their disease is metastatic to the liver. The liver metastatic disease should be confirmed cytologically or histologically at the time of study biopsy or prior to the study biopsy. All pre-study scans documenting disease must be done < 4 weeks prior to registration.
* Patients must have had no prior treatment with either irinotecan or oxaliplatin.
* Prior adjuvant therapy with fluoropyrimidine is allowed.
* Prior radiotherapy is allowed, but patients should have measurable disease outside the radiation port and/or progressive disease within the previously radiated volume. In addition, it must be at least 2 weeks since administration of radiation therapy and all signs of toxicity must have abated.
* Patients must have adequate renal and hepatic function (creatinine < 1.6 and calculated creatinine clearance [Cockcroft-Gault equation] > 60 ml/min; bilirubin < 2.0; and serum glutamic oxaloacetic transaminase [SGOT] less than 3 x normal limits) obtained within 4 weeks prior to registration.
* Alkaline phosphatase < 2.5 x upper normal limit (or < 5 x upper normal limit in the case of liver metastases or < 10 x upper normal limit in the case of bone disease)
* Patients must have absolute neutrophil count (ANC) > 1500/mm³ and platelet count > 100,000/mm³ within 4 weeks prior to registration.
* Have a negative serum or urine pregnancy test within 7 days prior to starting therapy (female patients of childbearing potential)

Exclusion Criteria:

* Pregnant and breast-feeding women are excluded from the study because effects on the fetus are unknown and there may be a risk of increased fetal wastage.
* Women of childbearing potential with either a positive or no pregnancy test (serum or urine) at baseline. Women/men of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.) Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
* Serious, uncontrolled, concurrent infection(s). Patients must have no evidence of significant active infection (e.g., pneumonia, peritonitis, wound abscess, etc.) at time of study entry.
* Life expectancy < 3 months
* Any prior fluoropyrimidine therapy (unless given in an adjuvant setting and completed at least 6 months earlier)
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil or known dihydropyrimidine dehydrogenase (DPD) deficiency
* Treatment for other carcinomas within the last 5 years, except cured non-melanoma skin and treated in-situ cervical cancer
* Participation in any investigational drug study
* Clinically significant cardiac disease of New York Heart Association Class III or greater (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Evidence of central nervous system (CNS) metastases (unless CNS metastases have been stable for > 3 months) or history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation
* Major surgery, open biopsy, or significant trauma injury within 28 days prior to Day 0
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy
* Impaired renal function (estimated creatinine clearance < 60ml/min as calculated with Cockcroft-Gault equation
* Unwillingness to give written informed consent
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Urine protein: creatinine ratio > 1.0 at screening
* Blood pressure of > 150/100 mmHg
* Unstable angina
* Clinically significant peripheral vascular disease
* Arterial thrombotic events, stroke or transient ischemic attack (TIA) within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, MD, Principal Investigator — H. Lee Moffitt Cancer Center & Research Institute / University of South Florida
Locations (12):
- United States (12):
  - North Broward Medical Center, Deerfield Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Center for Cancer Care & Research - Watson Clinic, Lakeland, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Martin Memorial, Stuart, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Bay Area Oncology, Tampa, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Space Coast Medical Associates, Titusville, Florida
  - St. Joseph's Candler Health System, Savannah, Georgia
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska

REFERENCES:
- See also: H. Lee Moffitt Cancer Center & Research Institute Web Page — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | XELOX + Bevacizumab | XELIRI + Bevacizumab
Started | 34 | 31
Completed | 26 (26 Participants were evaluable.) | 20 (20 Participants were evaluable.)
Not Completed | 8 | 11
Not completed — Insufficient Data for Analysis | 6 | 11
Not completed — Screen Failure | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XELOX + Bevacizumab | XELIRI + Bevacizumab | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 16 | 13 | 29
Age, Continuous [Mean (Full Range); unit: years] | 62.5 [39 to 88] | 64 [38 to 82.5] | 63 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Per Treatment Arm, Per Tumor Tissue Response Classifier
Description: Investigators would develop tumor tissue classifiers to predict response to the XELOX arm or XELIRI arm; with gene expression profiles on 75 patients on each of 2 arms, construct 2 classifiers to distinguish responders (complete responses, partial responses, stable disease) from non-responders (progressive disease).
Time Frame: 30 Days After End of Treatment - Average of 6 Months
Population: Low accrual and early termination prevented us from performing the planned analysis. Too few patients had both clinical and microarray data.
Arm/Group | XELOX + Bevacizumab | XELIRI + Bevacizumab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants Per Treatment Arm, With Overall Survival (OS)
Description: Investigators planned to evaluate the overall survival of colorectal cancer (CRC) patients treated with XELOX + bevacizumab (Arm A) or XELIRI + bevacizumab (Arm B).
Time Frame: 30 Days After End of Treatment - Average of 6 Months
Population: as for outcome 1
Arm/Group | XELOX + Bevacizumab | XELIRI + Bevacizumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Review of Serious Adverse Events (SAEs) To assess the toxicity associated with Arms A and B. Response rates and toxicity rates for each arm were to be estimated and exact (using Casella's method) 95% confidence intervals for those proportions computed. With the anticipated 75 patients in each arm, these estimated proportions would have standard errors not exceeding 7%.
Time Frame: 30 Days After End of Treatment - Average of 6 Months
Population: All participants.
Measure: Number; unit: participants
Arm/Group | XELOX + Bevacizumab | XELIRI + Bevacizumab
Number analyzed (Participants) | 34 | 31
participants | 9 | 11

ADVERSE EVENTS:
Time Frame: 5 years, 5 months
Arm/Group | XELOX + Bevacizumab | XELIRI + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 9/34 | 11/31
Other Adverse Events (participants affected / at risk) | 0/34 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XELOX + Bevacizumab (N=34) | XELIRI + Bevacizumab (N=31)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1) — Also experienced pain
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — 1 on Arm A also experienced vomiting and dehydration
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bilirubin - hospitalized (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Choking incident while taking tablet (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Death due to disease progression - liver (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) — Also experienced vomiting and abdominal pain
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) — 2 in Arm A and 1 in Arm B also had vomiting. 2 in Arm B also had nausea.
Diarrhea - persistent (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9/L) (General disorders) | 1 (1) | 0 (0)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) — 2 in Arm A and 3 in Arm B also experienced vomiting. 2 in Arm B also experienced diarrhea.
Obstructing lesion of the colon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain - headache (General disorders) | 0 (0) | 1 (1)
Perforation, GI - Duodenum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3) — 2 in Arm A and 3 in Arm B also experienced nausea. 1 in Arm B also experienced diarrhea.

LIMITATIONS AND CAVEATS:
Study was Terminated early, not Completed. Study Drug now on the market. Due to slow accrual, too few patients who had both clinical and microarray data to perform the proposed analysis. 65 of 92 patients consented were assigned to treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No